CLINICAL TRIAL: NCT07081100
Title: Study on the Effect of Probiotics on Improving Gastrointestinal Function in Patients With Non-organic Gastrointestinal Dysfunction
Brief Title: Probiotics and Non-Organic Gastrointestinal Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WK20250716
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic group (Experimental)
  Interventions: Dietary Supplement: Probiotic group

INTERVENTIONS:
Dietary Supplement: Probiotic group — Participants took a freeze-dried probiotic powder every day, half an hour after a meal.

SUMMARY:
To verify the improvement of gastrointestinal function in patients with non-organic gastrointestinal dysfunction after 4 weeks of intervention with compound probiotics.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form and agree to participate in the study.
* Ability to complete the study according to the trial protocol requirements.
* Aged 18-65 years.
* Clinical diagnosis of non-organic gastrointestinal dysfunction (e.g., functional dyspepsia, functional constipation) without other serious organic diseases.

Exclusion Criteria:

* Use of drugs affecting intestinal flora (antibiotics, probiotics, intestinal mucosal protectants, herbal medicines, etc.) for >1 week within 1 month prior to screening.
* Short-term use of products with functions similar to the investigational product, which may interfere with result interpretation.
* Antibiotic use during the study period.
* History of severe systemic diseases or malignancies.
* Allergy to any ingredient in the compound probiotic freeze-dried powder used in the trial.
* Pregnancy, lactation, or plans for pregnancy in the near future.
* Inability to participate due to personal reasons.
* Other conditions deemed unsuitable by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of gastrointestinal function in study participants | 4 weeks
  The severity of gastrointestinal symptoms was assessed by the Gastrointestinal Symptom Rating Scale (GSRS). Each item is scored from 1 (no symptoms) to 7 (extremely severe symptoms. Higher scores indicate worse gastrointestinal dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Ninth People's Hospital Suzhou Ninth Hospital affiliated to Soochow University, Suzhou, Jiangsu, China